CLINICAL TRIAL: NCT06480071
Title: The Role of Nasal Breathing for Perfomance in Elite Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Johan Hellgren, Professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Dnr 2020-03808
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Breathing, Mouth
MeSH Terms: conditions — Mouth Breathing | interventions — Oxymetazoline; Nasal Sprays

STUDY DESIGN:
Intervention Model Description: The nasal mucosa was decongested with oxymetazoline nasal spray 0.5mg/ml 2 sprays eacg nostril to achieve maximum nasal decongestion and to investigate if this promotes the physical performance during heavey exercise.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nasal decongestion during exercise (Experimental): Nasal decongestion with oxymetazomin nasal spray 0.05% 2 sprays each nostril 10 minutes before the exercise test
  Interventions: Drug: Oxymetazoline, 0.05% Nasal Spray

INTERVENTIONS:
Drug: Oxymetazoline, 0.05% Nasal Spray — 2 sprays each nostril before the excercise test.

SUMMARY:
This study investigates the contribution of nasal breathing to the performance during aerobic and anaerobic heavy exercise in 12 male elite cyclists. In a ramp test on a mechanically braked cycle ergometer (Monark LT2, Varberg, Sweden) VO2 max, heart rate, respiratory frequency, intranasal geometry and nasal airflow resitance as well as blood lactate and glucose was measured at each step of the ramp test and after a maximum exhaust test. Nasal breathing was randomized to three sepratae tests, normal open nose, decongested nose with oxymetazoline 0.5mg/ml, 2 sprays each nostril and with a nose clip. The study showed that in the test with the nose clip, mean blood lactate was significantly lower.

DETAILED DESCRIPTION:
Exercise experiments will be performed on12 elite male cyclists/triathletes, 20-40 years of age. The subjects should have a VO2max of ≥65 ml/min/kg. The subjects will perform pre-tests determining VO2max according to standard techniques. Subjects will be recruited through local contacts at clubs for cyclists and triathletes. Subjects should not have any medication, no nasal symptoms/disease and no asthma and be non-smokers. Subjects will be included after informed consent. All subjects answer a respiratory and training questionnaire. In total, all participants will undergo four visits to the exercise lab (CHP): the first visit for characterisation (pre-test) and the following three visits will be the exercise trials in a randomized order. All visits will take approximately 2 hours.

Experimental trials Diet and Activity Before Testing Participants will be instructed to refrain from alcohol and asked not to perform vigorous exercise on the day before each experimental trial, to record their diet on the first of these days, and to repeat this diet on days before subsequent trials.

Test day procedures Following an overnight fast, participants will be instructed to consume 500 ml plain water upon wakening. Upon arrival at the laboratory (CHP), height and nude body mass will be recorded, and a blood sample (hB) and a urine sample will be collected. A pre-trial urine specific gravity (USG) ≤1.025 (Atago, Tokyo, Japan) will be considered as a euhydrated state. Body composition will be assessed at the first experimental trial by dual-energy X-ray absorptiometry (iDXA; GE Medical Systems, Madison, WI, USA). Total fat and lean mass will be analyzed using enCore software (version 16.10).

Visual analogue scale for nasal symptoms will be recorded. The nose will be examined with anterior rhinometry and with a nasal endoscope. Spirometry will be performed. Intranasal geometry and nasal airway resistance will be measured immediately before during and after the exercise test.

Following the anthropometric measurements, an incremental maximal laboratory test will be performed on a mechanically braked cycle ergometer (Monark LT2, Varberg, Sweden) adapted with a racing saddle, drop handlebars, and clip-in pedals. Initial workload will be set at 110 W and increased by 35 W every 6 min, with 2-min recovery intervals/data collection points between workloads. With assistance of a metronome, pedal rate will be kept constant at 75 rpm through the entire test. Testing will be continued until the participant no longer can maintain the required pedal rate. Heart rate (HR) will be recorded every 5 s throughout the test (Polar Electro OY, model S10i, Finland). Blood samples (Figure) will be obtained to determine blood lactate concentration ([Lac]) and glucose immediately after each completed workload. [Lac] values attained during the last workload will be considered to be maximal. Maximal power output (Wmax) will be determined as the highest workload the participant can maintain for a complete 6-min period. Environmental conditions during the experimental trials will be approximately 20°C and 40-50% relative humidity.

The exercise intensity corresponding to the onset of blood lactate accumulation (OBLA) will be identified on the [Lac]-power output curve by straight-line interpolation between the two closest points as the power output eliciting a [Lac] of 4 mmol/l . Power output and HR values at OBLA (W˙OBLA and HROBLA, respectively) will be determined by straight-line interpolation.

Outcomes VO2, CO2, HR, ventilation rate, ventilatory equivalents for oxygen and CO2 [Veq∙O2

-1 and Veq∙CO2-1], RPE, time to exhaustion, Aerobic and anaerobic threshold

ELIGIBILITY:
Inclusion Criteria:

* male subjects
* age 18-40
* elite cyclists or Triathlon athletes
* minimum VO2max of ≥65 ml/min/kg on pretest.

Exclusion Criteria:

* non-male
* <18>40 years of age
* non-elite cyclists or Triathlon athletes
* less than VO2max of ≥65 ml/min/kg on pretest

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — To increase standardisation regarding physical performance only one sex was included in the study
Enrollment: 12 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
VO2 max | 7 minutes per cycle
  maximum oxygen upptake during exrecise
blood lactate | 7 minutes per cycle
  lactic acid, a cmponent produced during anaerobic heavy exercise
Effect | 7 minutes per cycle
  Watt effect generated during exercise

SECONDARY OUTCOMES:
HR | 7 minutes per cycle
  heart rate per minute
nasal air flow resistance | 7 minutes per cycle
  nasal patency

CONTACTS AND LOCATIONS:
Overall Officials: Johan Hellgren, MD, PhD, Professor, Principal Investigator — Department of ENT Sahlgrenska University Hospital Sweden
Locations (1):
- Department of ENT Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No